CLINICAL TRIAL: NCT05366725
Title: A MULTI-CENTRE NON-INTERVENTIONAL STUDY TO DESCRIBE THE EARLY CLINICAL EXPERIENCE OF AVELUMAB USED AS MONOTHERAPY FOR THE FIRST-LINE MAINTENANCE TREATMENT OF ADULT PATIENTS WITH LOCALLY ADVANCED OR METASTATIC UROTHELIAL CARCINOMA WHO ARE PROGRESSION-FREE FOLLOWING PLATINUM-BASED CHEMOTHERAPY
Brief Title: A Study to Learn About the Study Medicine (Called Avelumab) in People With Advanced Urothelial Cancer After Chemotherapy
Status: Completed | Type: Observational
Sponsor: Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Other Study IDs: B9991047
Record Dates: First submitted 2022-05-04; First posted 2022-05-09 (Actual); Results first posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Urothelial Cancer
MeSH Terms: interventions — avelumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other

GROUPS / COHORTS (1):
- Adult patients with locally advanced or metastatic urothelial cancer
  Interventions: Drug: Avelumab

INTERVENTIONS:
Drug: Avelumab — As provided in real world practice

SUMMARY:
The purpose of this clinical trial is to learn about the safety and effects of the study medicine (called Avelumab) in people with advanced urothelial (bladder) cancer (UC) whose disease hasn't worsened after receiving chemotherapy.

This study is seeking participants who:

1. Have UC that cannot be operated on or has spread to other parts of the body
2. Received 1st line platinum-based chemotherapy and had stable disease, partial response, or complete response to this treatment
3. Received Avelumab as indicated as the only therapy for the first-line maintenance who are progression-free following platinum-based chemotherapy
4. Are 18 years or older on the date that they start taking Avelumab

All participants in this study will receive Avelumab, a standard treatment for urothelial carcinoma. Participants will take part in this study for about 4 years. During this time, they will take Avelumab as instructed in the real-world setting. We will study the experiences of people receiving the study medicine. This will help us decide if the study medicine is safe and effective.

DETAILED DESCRIPTION:
The primary objective of this study is to estimate real-world overall survival (rwOS) in a real-world cohort of patients treated with avelumab monotherapy for the first-line maintenance treatment of adult patients with locally advanced or metastatic UC who are progression-free following platinum-based chemotherapy.

The secondary objectives are:

1. To describe the clinical and demographic characteristics of the study population
2. To estimate real-world progression-free survival (rwPFS)
3. To describe treatment characteristics of 1L anti-cancer therapies received prior to the initiation of avelumab as 1Lmaintenance therapy
4. To describe treatment patterns after initiation of avelumab as 1L maintenance therapy
5. To describe the adverse events (AEs) explicitly attributed to avelumab in a real-world population
6. To describe real-world all-cause associated healthcare resource burden associated with avelumab therapy

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a diagnosis of locally advanced or metastatic UC, either de novo or relapsed
2. Patients received 1L platinum-based chemotherapy and had stable disease, partial response, or complete response to this treatment
3. Patients received avelumab as indicated as a monotherapy for the first-line maintenance treatment of adult patients with locally advanced or metastatic UC who are progression-free following platinum-based chemotherapy
4. Patients aged ≥18 years on the date that they commenced avelumab -

Exclusion Criteria:

1. Patients whose hospital records are not available for review
2. Patients who are receiving an investigational medicinal product as part of a clinical trial at the time of maintenance therapy with avelumab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with a diagnosis of locally advanced or metastatic UC, either de novo or relapsed who are progression-free following completion of platinum-based chemotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2022-06-29 (Actual); Primary Completion 2024-06-27 (Actual); Study Completion 2024-06-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany
Locations (10):
- United Kingdom (10):
  - University Hospitals Bristol, Bristol
  - Beatson West of Scotland Cancer Centre, Glasgow
  - Royal Surrey County Hospital, Guildford
  - University College London Hospital, London
  - Guy's and St Thomas' Hospital, London
  - The Christie NHS Foundation Trust, Manchester
  - Clatterbridge Hospital, Metropolitan Borough of Wirral
  - Churchill Hospital, Oxford
  - Royal Preston Hospital, Preston
  - Lister Hospital, Stevenage

IPD SHARING:
Plan to Share IPD: No
We are committed to enhancing public health through responsible sharing of clinical trial data. Following approval of a new product or a new indication for an approved product in both the US and the European Union, the study sponsor and/or its affiliated companies will share study protocols, anonymized patient data and study level data, and redacted clinical study reports with qualified scientific and medical researchers, upon request, as necessary for conducting legitimate research. Further information on how to request data can be found on our website bit.ly/IPD21

REFERENCES:
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en/trial-details/?id=B9991047
- See also: Medical Information Location Map - Med Info Contacts — https://www.merckgroup.com/en/company/contact-us/medinfo-contact-map.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Participants With Locally Advanced or Metastatic Urothelial Cancer (UC): Participants with locally advanced or metastatic UC whose disease has not progressed following first line platinum-based chemotherapy and were treated with avelumab as a first line maintenance therapy were enrolled in this study. No intervention was administered and only clinical data collected in routine clinical care was accessed and analyzed as part of this noninterventional study. Data was extracted from participants medical records and hospital charts.
Period: Overall Study
Arm/Group | Participants With Locally Advanced or Metastatic Urothelial Cancer (UC)
Started | 106
Completed | 106
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Participants With Locally Advanced or Metastatic Urothelial Cancer (UC): Participants with locally advanced or metastatic UC whose disease has not progressed following first line platinum-based chemotherapy and were treated with avelumab as a first line maintenance therapy were enrolled in this study. No intervention was administered and only clinical data collected in routine clinical care was accessed and analyzed as part of this noninterventional study. Data was extracted from patient medical records and hospital charts.
Arm/Group | Participants With Locally Advanced or Metastatic Urothelial Cancer (UC)
Number analyzed (Participants) | 106
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.5 (12.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 78
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 106

OUTCOME MEASURES:

1. Primary Outcome: Real-World Overall Survival
Description: Real-World Overall Survival is the time from participant eCRF index date (avelumab initiation between September 2020 to November 2021) to date of death by any cause, or date of censoring, inclusive of start and end date. Analysis was performed using Kaplan-Meier method.
Time Frame: From participant eCRF index date (avelumab initiation between September 2020 to November 2021) to date of death by any cause, or date of censoring (whichever is first) (up to 24-months from initiation of avelumab treatment)
Population: The Full Analysis Set comprised of participants who met the inclusion criteria and did not meet the exclusion criteria.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Participants With Locally Advanced or Metastatic Urothelial Cancer (UC)
Number analyzed (Participants) | 106
months | 16.8 [11.6 to 23.4]

2. Secondary Outcome: Clinical Characteristics: Time From First Diagnosis to Locally Advanced or Metastatic Diagnosis
Description: Time from First Diagnosis to Locally Advanced or Metastatic Diagnosis is the time between date of first diagnosis and date of locally advanced or metastatic diagnosis. Due to retrospective nature of study, the diagnosis data was collected retrospectively before participants were enrolled into the study, hence timeframe exceeds the study duration in this outcome measure.
Time Frame: Time between date of first diagnosis and date of locally advanced or metastatic diagnosis measured at baseline (date of locally advanced or metastatic diagnosis) (Up to 621.4 weeks)
Population: The Full Analysis Set comprised of participants who met the inclusion criteria and did not meet the exclusion criteria.
Measure: Median (Full Range); unit: weeks
Arm/Group | Participants With Locally Advanced or Metastatic Urothelial Cancer (UC)
Number analyzed (Participants) | 106
weeks | 67.4 [0.0 to 621.4]

3. Secondary Outcome: Clinical Characteristics: Participant's Age at Locally Advanced or Metastatic Diagnosis
Description: Age (in years) at date of locally advanced or metastatic cancer diagnosis. Calculated as the number of years between date of birth and date of locally advanced or metastatic diagnosis, rounded down to the nearest whole year of age was reported. Due to retrospective nature of study, the diagnosis data was collected retrospectively before participants were enrolled into the study, hence timeframe exceeds the study duration in this outcome measure.
Time Frame: as for outcome 2
Population: The Full Analysis Set comprised of participants who met the inclusion criteria and did not meet the exclusion criteria.
Measure: Mean (Standard Deviation); unit: years
Arm/Group | Participants With Locally Advanced or Metastatic Urothelial Cancer (UC)
Number analyzed (Participants) | 106
years | 68.5 (11.46)

4. Secondary Outcome: Clinical Characteristics: Participant's Stage of UC at Locally Advanced or Metastatic Diagnosis
Description: The Stage of UC of participants at Locally Advanced or Metastatic Diagnosis was reported as recorded in eCRF Q13: Stage IIIA, Stage IIIB, Stage IVA or Stage IVB. Urothelial cancer stages III to IVB indicate progressive spread of the disease. In Stage IIIA, the cancer has invaded nearby tissues like the prostate, uterus, or vagina, or has reached one lymph node in the pelvis. Stage IIIB involves spread to two or more lymph nodes in that region. In Stage IVA, the cancer extends further to nearby organs such as the pelvic or abdominal wall, or to distant lymph nodes. Stage IVB represents the most advanced stage, where the cancer has metastasized to distant organs like the lungs, liver, or bones. Due to retrospective nature of study, the diagnosis data was collected retrospectively before participants were enrolled into the study, hence timeframe exceeds the study duration in this outcome measure.
Time Frame: as for outcome 2
Population: The Full Analysis Set comprised of participants who met the inclusion criteria and did not meet the exclusion criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Locally Advanced or Metastatic Urothelial Cancer (UC)
Number analyzed (Participants) | 106
Participants
  Stage IIIA | 13
  Stage IIIB | 8
  Stage IVA | 20
  Stage IVB | 55
  Unknown | 10

5. Secondary Outcome: Clinical Characteristics: Participant's Histology at Locally Advanced or Metastatic Diagnosis
Description: Participant's Histology at Locally Advanced or Metastatic Diagnosis was reported. Number of participants with histology of Pure urothelial cancer, mixed urothelial with component of another pathology, or other were reported. Due to retrospective nature of study, the diagnosis data was collected retrospectively before participants were enrolled into the study, hence timeframe exceeds the study duration in this outcome measure.
Time Frame: as for outcome 2
Population: The Full Analysis Set comprised of participants who met the inclusion criteria and did not meet the exclusion criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Locally Advanced or Metastatic Urothelial Cancer (UC)
Number analyzed (Participants) | 106
Participants
  Pure urothelial cancer (transitional cell carcinoma) | 86
  Mixed urothelial with component of another pathology | 11
  Other | 9

6. Secondary Outcome: Clinical Characteristics: Number of Participants With De Novo Disease or Newly Relapsed at Locally Advanced or Metastatic Diagnosis
Description: Number of participants with de novo disease or newly relapsed at locally advanced or metastatic diagnosis was reported. Due to retrospective nature of study, the diagnosis data was collected retrospectively before participants were enrolled into the study, hence timeframe exceeds the study duration in this outcome measure.
Time Frame: as for outcome 2
Population: The Full Analysis Set comprised of participants who met the inclusion criteria and did not meet the exclusion criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Locally Advanced or Metastatic Urothelial Cancer (UC)
Number analyzed (Participants) | 106
Participants
  De novo disease | 59
  Newly relapsed | 46
  Unknown | 1

7. Secondary Outcome: Clinical Characteristics: Participant's Programmed Death-Ligand 1 (PD-L1) Tumour Assessment Immune Cell (IC) Test Result at Locally Advanced or Metastatic Diagnosis
Description: Participants PD-L1 tumour assessment immune cell (IC) test result at Locally Advanced or Metastatic Diagnosis was reported. Due to retrospective nature of study, the diagnosis data was collected retrospectively before participants were enrolled into the study, hence timeframe exceeds the study duration in this outcome measure.
Time Frame: as for outcome 2
Population: The Full Analysis Set comprised of participants who met the inclusion criteria and did not meet the exclusion criteria.
Measure: Mean (Standard Deviation); unit: cubic/millimeter (mm) 3
Arm/Group | Participants With Locally Advanced or Metastatic Urothelial Cancer (UC)
Number analyzed (Participants) | 106
cubic/millimeter (mm) 3 | 2.0 (2.45)

8. Secondary Outcome: Clinical Characteristics: Number of Participants With Eastern Cooperative Oncology Group (ECOG) Performance Status Score of 0, 1 and 2, 3 or 4
Description: ECOG-PS assessed participant's performance status on a 5 point scale: 0= fully active/able to carry on all pre-disease activities without restriction; 1= restricted in physically strenuous activity, ambulatory/able to carry out light or sedentary work; 2= ambulatory (>50% of waking hours), capable of all self-care, unable to carry out any work activities; 3= capable of only limited self-care, confined to bed/chair >50% of waking hours; 4= completely disabled, cannot carry on any self-care, totally confined to bed/chair. Due to retrospective nature of study, the diagnosis data was collected retrospectively before participants were enrolled into the study, hence timeframe exceeds the study duration in this outcome measure.
Time Frame: as for outcome 2
Population: The Full Analysis Set comprised of participants who met the inclusion criteria and did not meet the exclusion criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Locally Advanced or Metastatic Urothelial Cancer (UC)
Number analyzed (Participants) | 106
Participants
  0 | 35
  1 | 36
  2, 3, or 4 | 5
  Not recorded | 30

9. Secondary Outcome: Clinical Characteristics: Participants Site of Metastases
Description: Participants site of metastases: Lymph nodes, Bone, Lung, Liver, Peritoneum or other was reported. Participants could have one or more sites of metastases. Due to retrospective nature of study, the diagnosis data was collected retrospectively before participants were enrolled into the study, hence timeframe exceeds the study duration in this outcome measure.
Time Frame: as for outcome 2
Population: The Full Analysis Set comprised of participants who met the inclusion criteria and did not meet the exclusion criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Locally Advanced or Metastatic Urothelial Cancer (UC)
Number analyzed (Participants) | 106
Participants
  Lymph nodes | 64
  Bone | 21
  Lung | 32
  Liver | 18
  Other | 19

10. Secondary Outcome: Clinical Characteristics: Number of Participants With Prior Radical Treatment of Primary UC at Locally Advanced or Metastatic Diagnosis
Description: The number of participants with prior radical treatment of primary UC at Locally Advanced or Metastatic Diagnosis were reported. Due to retrospective nature of study, the diagnosis data was collected retrospectively before participants were enrolled into the study, hence timeframe exceeds the study duration in this outcome measure.
Time Frame: as for outcome 2
Population: The Full Analysis Set comprised of participants who met the inclusion criteria and did not meet the exclusion criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Locally Advanced or Metastatic Urothelial Cancer (UC)
Number analyzed (Participants) | 106
Participants
  Yes | 47
  No | 57
  Unknown | 2

11. Secondary Outcome: Clinical Characteristics: Number of Participants With Prior Adjuvant or Neoadjuvant System Therapy at Locally Advanced or Metastatic Diagnosis
Description: The number of participants with prior adjuvant or neoadjuvant system therapy at Locally Advanced or Metastatic Diagnosis were reported. Due to retrospective nature of study, the diagnosis data was collected retrospectively before participants were enrolled into the study, hence timeframe exceeds the study duration in this outcome measure.
Time Frame: as for outcome 2
Population: The Full Analysis Set comprised of participants who met the inclusion criteria and did not meet the exclusion criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Locally Advanced or Metastatic Urothelial Cancer (UC)
Number analyzed (Participants) | 106
Participants
  Yes | 35
  No | 69
  Unknown | 2

12. Secondary Outcome: Age of Participants at Avelumab Initiation
Description: The age of participants at avelumab initiation was reported.
Time Frame: At Index date (date of avelumab initiation between September 2020 to November 2021 ) as reported in the eCRF.
Population: The Full Analysis Set comprised of participants who met the inclusion criteria and did not meet the exclusion criteria.
Measure: Mean (Standard Deviation); unit: years
Arm/Group | Participants With Locally Advanced or Metastatic Urothelial Cancer (UC)
Number analyzed (Participants) | 106
years | 69.3 (11.41)

13. Secondary Outcome: Real-World Progression-Free Survival (Rw-PFS)
Description: Rw-PFS is the time from the start date of avelumab treatment to the first date of either: any evidence of progression or date of death.
Time Frame: as for outcome 1
Population: The Full Analysis Set comprised of participants who met the inclusion criteria and did not meet the exclusion criteria.
Measure: Median (Full Range); unit: months
Arm/Group | Participants With Locally Advanced or Metastatic Urothelial Cancer (UC)
Number analyzed (Participants) | 106
months | 8.7 [7.1 to 14.2]

14. Secondary Outcome: Treatment Characteristics: Type of First Systemic Anticancer Treatment (SACT) Regimen Received Before Avelumab Start Date
Description: Number of participants who received type of First SACT regimen received were reported.
Time Frame: From date of locally advanced or metastatic diagnosis to index date (Day 0) (avelumab initiation date between Sep 2020 to Nov 2021 as reported in the eCRF) (Up to 24 months)
Population: The Full Analysis Set comprised of participants who met the inclusion criteria and did not meet the exclusion criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Locally Advanced or Metastatic Urothelial Cancer (UC)
Number analyzed (Participants) | 106
Participants
  Cisplatin/gemcitabine | 49
  Carboplatin/gemcitabine | 55
  Unknown | 2

15. Secondary Outcome: Treatment Characteristics: Number of First- Line Systematic Anti-Cancer Therapy (SACT) Cycles Received
Description: Number of first line SACT cycles received by participants was reported as treatment characteristics.
Time Frame: as for outcome 14
Population: The Full Analysis Set comprised of participants who met the inclusion criteria and did not meet the exclusion criteria.
Measure: Mean (Standard Deviation); unit: cycles
Arm/Group | Participants With Locally Advanced or Metastatic Urothelial Cancer (UC)
Number analyzed (Participants) | 106
cycles | 5.3 (1.16)

16. Secondary Outcome: Treatment Characteristics: Number of Participants Switching Between Different Platinum-Based Chemotherapies
Description: Number of participants switching between different platinum-based chemotherapies were reported.
Time Frame: as for outcome 14
Population: The Full Analysis Set comprised of participants who met the inclusion criteria and did not meet the exclusion criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Locally Advanced or Metastatic Urothelial Cancer (UC)
Number analyzed (Participants) | 106
Participants
  Yes | 7
  No | 99

17. Secondary Outcome: Treatment Characteristics: Time From Completion of First Line Systematic Anti-Cancer Therapy (SACT) to Start of Avelumab
Description: Time from completion of first line SACT to start of avelumab was reported. Calculated as the number of days from the end date of the last first line SACT cycle to the start date of avelumab, inclusive of the start and end dates of this period.
Time Frame: From date of the last record of first line SACT to index date (Day 0) (avelumab initiation date between September 2020 - November 2021 as reported in the eCRF) (Up to 24 months)
Population: The Full Analysis Set comprised of participants who met the inclusion criteria and did not meet the exclusion criteria.
Measure: Median (Full Range); unit: weeks
Arm/Group | Participants With Locally Advanced or Metastatic Urothelial Cancer (UC)
Number analyzed (Participants) | 106
weeks | 8.5 [0.43 to 26.1]

18. Secondary Outcome: Treatment Characteristics: Response to First Line Therapy
Description: Response to first line therapy was reported. Response to first line SACT as reported in eCRF included: Complete Response (CR), Partial Response (PR) and Stable disease. The definitions of tumor responses are as follows: Complete or PR as the best adjudication result (CR > PR > stable disease [SD] > progressive disease [PD]) complies with the RECIST tumor assessment guidelines as closely as possible in clinical practice.
Time Frame: From date of first line SACT initiation to index date (Day 0) (avelumab initiation date between September 2020 - November 2021 as reported in the eCRF) (Up to 24 months)
Population: The Full Analysis Set comprised of participants who met the inclusion criteria and did not meet the exclusion criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Locally Advanced or Metastatic Urothelial Cancer (UC)
Number analyzed (Participants) | 106
Participants
  Complete response | 9
  Partial response | 54
  Stable disease | 42
  Unknown | 1

19. Secondary Outcome: Treatment Characteristics: Response to First-Line Therapy Based on Computed Tomography (CT) Scan Evidence
Description: Response to First Line therapy based on CT scan evidence was reported. Response to first line SACT was judged based on CT scan evidence after the last cycle of first line SACT, as reported in eCRF. Reported as Yes or No.
Time Frame: as for outcome 18
Population: The Full Analysis Set comprised of participants who met the inclusion criteria and did not meet the exclusion criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Locally Advanced or Metastatic Urothelial Cancer (UC)
Number analyzed (Participants) | 106
Participants
  Yes | 101
  No | 5

20. Secondary Outcome: Treatment Patterns: Duration of Treatment With Avelumab
Description: Duration was derived based on the date of avelumab initiation and the last date of avelumab treatment.
Time Frame: From (avelumab initiation date between September 2020 - November 2021 as reported in the eCRF) to end date of avelumab, or date of censoring (whichever is first), assessed upto 24 months after avelumab initiation
Population: The Full Analysis Set comprised of participants who met the inclusion criteria and did not meet the exclusion criteria.
Measure: Median (Full Range); unit: weeks
Arm/Group | Participants With Locally Advanced or Metastatic Urothelial Cancer (UC)
Number analyzed (Participants) | 106
weeks | 34.2 [0.14 to 104.6]

21. Secondary Outcome: Treatment Patterns: Number of Participants Who Received Second-Line Therapy as Per eCRF
Description: Number of participants who received second-line therapy were reported.
Time Frame: From (avelumab initiation date between September 2020 - November 2021 as reported in the eCRF) and end of follow-up (upto 24 months after avelumab initiation)
Population: The Full Analysis Set comprised of participants who met the inclusion criteria and did not meet the exclusion criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Locally Advanced or Metastatic Urothelial Cancer (UC)
Number analyzed (Participants) | 106
Participants | 15

22. Secondary Outcome: Treatment Patterns: Time Interval Between Start of Avelumab and Start of Second-Line Therapy
Description: Time interval was derived using the dates of avelumab initiation and initiation of first regimen of second line therapy. This parameter was calculated only among participants who go on to receive second-line therapy after avelumab initiation.
Time Frame: From (avelumab initiation date between September 2020 - November 2021 as reported in the eCRF)to start of second-line therapy assessed upto 24 months after avelumab initiation.
Population: The Full Analysis Set comprised of participants who met the inclusion criteria and did not meet the exclusion criteria.
Measure: Median (Full Range); unit: weeks
Arm/Group | Participants With Locally Advanced or Metastatic Urothelial Cancer (UC)
Number analyzed (Participants) | 106
weeks | 38.7 [9.1 to 92.0]

23. Secondary Outcome: Treatment Patterns: Systematic Anti-Cancer Therapy Regimen Received as Second Line Therapy
Description: Number of participants who received Systematic Anti-Cancer Therapy Regimen as Second Line Therapy was reported.
Time Frame: From avelumab initiation date between September 2020 - November 2021 as reported in the eCRF and upto 24 months after avelumab initiation
Population: The Full Analysis Set comprised of participants who met the inclusion criteria and did not meet the exclusion criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Locally Advanced or Metastatic Urothelial Cancer (UC)
Number analyzed (Participants) | 106
Participants | 5 [9.1 to 92.0]

24. Secondary Outcome: Treatment Patterns: High Dose Systemic Steroid Use
Description: Number of participants with high dose systemic steroid use was reported.
Time Frame: From avelumab initiation date between September 2020 - November 2021 as reported in the eCRF up to 24 months after avelumab initiation
Population: The Full Analysis Set comprised of participants who met the inclusion criteria and did not meet the exclusion criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Locally Advanced or Metastatic Urothelial Cancer (UC)
Number analyzed (Participants) | 106
Participants
  Yes | 24
  No | 80
  Unknown | 2

25. Secondary Outcome: Number of Participants With Adverse Events (AEs) Explicitly Attributed to Avelumab in a Real-World Population
Description: The number of separate AEs recorded per participants (with explicit linkage in the medical notes to avelumab) will be calculated using data from eCRF (each reported event on the eCRF counts as a separate AE).
Time Frame: as for outcome 1
Population: The Full Analysis Set comprised of participants who met the inclusion criteria and did not meet the exclusion criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Locally Advanced or Metastatic Urothelial Cancer (UC)
Number analyzed (Participants) | 106
Participants | 80

26. Secondary Outcome: Healthcare Resource Burden Associated With Avelumab Therapy: Accident and Emergency Visits
Description: The number of accident and emergency visits recorded per participant as reported on the eCRF was used to calculate the rate of events per participant per year of follow-up time.
Time Frame: as for outcome 1
Population: The Full Analysis Set comprised of participants who met the inclusion criteria and did not meet the exclusion criteria.
Measure: Mean (Standard Deviation); unit: number of accident&emergency visits/year
Arm/Group | Participants With Locally Advanced or Metastatic Urothelial Cancer (UC)
Number analyzed (Participants) | 106
number of accident&emergency visits/year | 1.9 (1.67)

27. Secondary Outcome: Healthcare Resource Burden Associated With Avelumab Therapy: Hospitalizations
Description: The number of hospital admissions recorded per participant as reported on the eCRF was used to calculate the rate of events per participant per year of follow-up time
Time Frame: From participant electronic case report form (eCRF) index date (avelumab initiation between September 2020 to November 2021) to date of death by any cause, or date of censoring (whichever is first) (up to 24-months from initiation of avelumab treatment)
Population: The Full Analysis Set comprised of participants who met the inclusion criteria and did not meet the exclusion criteria.
Measure: Mean (Standard Deviation); unit: rate of hospitalization per year
Arm/Group | Participants With Locally Advanced or Metastatic Urothelial Cancer (UC)
Number analyzed (Participants) | 106
rate of hospitalization per year | 2.7 (3.81)

28. Secondary Outcome: Healthcare Resource Burden Associated With Avelumab Therapy: Participants Duration of Hospitalisation
Description: Duration of Hospitalisation was reported.
Time Frame: Time from the start date of platinum-basedchemotherapeutic treatment to the earliest of date of death or date of censoring,as reported on the eCRF assessed up to 24 months from avelumab initiation (index date)
Population: The Full Analysis Set comprised of participants who met the inclusion criteria and did not meet the exclusion criteria.
Measure: Median (Full Range); unit: days
Arm/Group | Participants With Locally Advanced or Metastatic Urothelial Cancer (UC)
Number analyzed (Participants) | 106
days | 14.5 [0.5 to 172.3]

29. Secondary Outcome: Real-World Overall Survival
Description: Real world overall suvival was the time from the start date of platinum-based chemotherapeutic treatment to the earliest of date of death or date of censoring, as reported on the eCRF.
Time Frame: as for outcome 27
Population: The Full Analysis Set comprised of participants who met the inclusion criteria and did not meet the exclusion criteria.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Participants With Locally Advanced or Metastatic Urothelial Cancer (UC)
Number analyzed (Participants) | 106
months | 21.8 [17.0 to 28.9]

ADVERSE EVENTS:
Time Frame: Up to 24-months from initiation of avelumab treatment
Description: The Full Analysis Set comprised of participants who met the inclusion criteria and did not meet the exclusion criteria.
Arm/Group | Participants With Locally Advanced or Metastatic Urothelial Cancer (UC)
All-Cause Mortality (participants affected / at risk) | 66/106
Serious Adverse Events (participants affected / at risk) | 34/106
Other Adverse Events (participants affected / at risk) | 78/106
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Participants With Locally Advanced or Metastatic Urothelial Cancer (UC) (N=106)
Disease progression (General disorders) | 11
Pneumonitis (Infections and infestations) | 3
Dermatitis (Skin and subcutaneous tissue disorders) | 2
Infusion reaction (General disorders) | 2
Diabetes Mellitus (Endocrine disorders) | 1
Sub-dural Hemorrhage (Nervous system disorders) | 1
Pain (General disorders) | 1
Immunotherapy induced Encephalitis (Nervous system disorders) | 1
Incidental acute kidney injury (Renal and urinary disorders) | 1
Skin reaction (Skin and subcutaneous tissue disorders) | 1
Hypersensitivity (Immune system disorders) | 1
Deranged Liver Function Tests (Hepatobiliary disorders) | 1
Lack of efficacy (General disorders) | 1
Myositis (Musculoskeletal and connective tissue disorders) | 1
Vestibular neuritis (Nervous system disorders) | 1
Left Flank Pain (General disorders) | 1
Febrile Neutropenia (Blood and lymphatic system disorders) | 1
Hypophosphatemia (Investigations) | 1
Metastatic Spinal Cord Compression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Bone Metastases (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Participants With Locally Advanced or Metastatic Urothelial Cancer (UC) (N=106)
Disease progression (General disorders) | 28
Lack of efficacy (General disorders) | 14
Fatigue (General disorders) | 11
Rash (Skin and subcutaneous tissue disorders) | 8
Nephritis (Renal and urinary disorders) | 5
Hypothyroidism (Endocrine disorders) | 9
Transaminitis (Hepatobiliary disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 4
Toxicity (General disorders) | 2
Diarrhea (Gastrointestinal disorders) | 4
Vomiting (Gastrointestinal disorders) | 2
Myositis (Musculoskeletal and connective tissue disorders) | 1
Constipation (Gastrointestinal disorders) | 2
Hyperthyroidism (Endocrine disorders) | 1
Hepatitis (Hepatobiliary disorders) | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 2
Lichenoid drug eruption (Skin and subcutaneous tissue disorders) | 1
Itch and macular rash (Skin and subcutaneous tissue disorders) | 2
Infusion reaction (General disorders) | 2
Rash and balanitis (Skin and subcutaneous tissue disorders) | 1
Palmar-plantar erythema (Skin and subcutaneous tissue disorders) | 1
Loss of appetite (Gastrointestinal disorders) | 1
Itch and maculopustular rash (Skin and subcutaneous tissue disorders) | 1
Low Cortisol (Endocrine disorders) | 1
Adrenal insufficiency (Endocrine disorders) | 2
Urticaria (Skin and subcutaneous tissue disorders) | 1
Skin rash in forehead (Skin and subcutaneous tissue disorders) | 1
Itch scalp (Skin and subcutaneous tissue disorders) | 1
Bone metastases (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Residual neuropathy (Nervous system disorders) | 1
Papular rash on legs (Skin and subcutaneous tissue disorders) | 1
Fevers and chills (General disorders) | 1
ALT increased (Hepatobiliary disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Sequelae (General disorders) | 1
Anorexia (Psychiatric disorders) | 1
Acute Kidney Injury (Renal and urinary disorders) | 1
Creatinine Increased (Renal and urinary disorders) | 2
Urinary Tract Infection (Infections and infestations) | 1
Pneumonitis (Infections and infestations) | 1
Hypersensitivity reaction (Immune system disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Abdominal Pain (Gastrointestinal disorders) | 1
Hypomagnesemia (Investigations) | 1
Hypocalcemia (Investigations) | 1
Neutropenia (Investigations) | 1
Pelvic Pain (Gastrointestinal disorders) | 1
Urinary Symptoms (Renal and urinary disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Neuropathy (Nervous system disorders) | 1
Sore mouth (Gastrointestinal disorders) | 1
Itchy skin (Skin and subcutaneous tissue disorders) | 2
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1
Folliculitis (Skin and subcutaneous tissue disorders) | 2
Peripheral oedema (Vascular disorders) | 1
Itching (Skin and subcutaneous tissue disorders) | 2
Maculopapular Rash (Skin and subcutaneous tissue disorders) | 3
Immune related transaminitis (Hepatobiliary disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2023-07-03): https://cdn.clinicaltrials.gov/large-docs/25/NCT05366725/Prot_000.pdf
  • Statistical Analysis Plan (2021-12-01): https://cdn.clinicaltrials.gov/large-docs/25/NCT05366725/SAP_001.pdf